CLINICAL TRIAL: NCT00496288
Title: Phase II Multicenter Clinical Trial of Prophylactic Irradiation to the Contralateral Breast for BRCA Mutation Carriers Undergoing Treatment for Breast Cancer
Brief Title: Prophylactic Irradiation to the Contralateral Breast for BRCA Mutation Carriers Undergoing Treatment for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Rambam Health Care Campus (Other); Tel-Aviv Sourasky Medical Center (Other Government); Sheba Medical Center (Other Government); Soroka University Medical Center (Other); Western Galilee Hospital-Nahariya (Other Government); Rabin Medical Center (Other)
Responsible Party: Ella Evron, MD, Assaf-Harofeh Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102/07 (HT4351)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2008-06

CONDITIONS: Breast Cancer
Keywords: BRCA mutation; Breast cancer; Prophylactic breast irradiation; Prevention of contralateral breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prophylactic irradiation (Experimental): prophylactic contralateral breast irradiation
  Interventions: Radiation: Prophylactic radiation to the contralateral breast
- controls (No Intervention): Those that do not opt for prophylactic irradiation or mastectomy

INTERVENTIONS:
Radiation: Prophylactic radiation to the contralateral breast — The contralateral breast will be treated with 2 tangent fields, using 1.8-2 Gy/fx to a total dose of 50-50.4 Gy. The whole breast will be treated according to traditional guidelines and as described in the RTOG/NSABP B39 study. The heart should be maximally blocked for left sided breasts, included lung tissue should be reduced to minimum. No overlapping field is allowed on the skin between the two breast fields in the midline. Maximal dose should not exceed 110%
  Arms: prophylactic irradiation

SUMMARY:
Women with BRCA germline mutations face a very high risk of developing breast cancer during their lives. It was shown that for carrier patients, breast conservation, comprising of lumpectomy followed by whole breast radiation, was not associated with increased risk of ipsilateral breast cancer recurrence as compared with non carriers (10-15% over 10 years), especially if they also underwent prophylactic oophorectomy. Yet their risk of subsequent contralateral breast cancer was significantly increased, reported as high as 25-30% over 10 years and 40% over 15 years, as compared to 3% and 7% respectively in non carriers. The reduction in ipsilateral disease was attributed to radiation of the affected breast. We propose that for breast cancer patients with BRCA germline mutation that choose to have breast-conserving therapy and refuse prophylactic contralateral mastectomy, prophylactic radiation to the contralateral breast may reduce the rate of subsequent contralateral breast cancer and offer an option for risk reduction.

DETAILED DESCRIPTION:
Trial design and statistics:

This is a multi center- phase II open comparative trial. "Patients" - Those who choose prophylactic contralateral breast irradiation. "Controls" - Those that do not opt for prophylactic irradiation or mastectomy. Objective - to compare the rate of contralateral breast cancer in "patients" versus "controls".

Assuming that 2/3 of the eligible carrier breast cancer patients refuse the procedure: To detect a difference of 10% vs. 25% in the incidence of contralateral breast cancer with power = 80%, alpha = 0.05, 80 patients and 160 controls need to be enrolled.

Treatment:

Chemotherapy, Hormonal therapy and XRT to the affected breast as per treating institution.

Radiation therapy:

Patients will undergo a pre-treatment planning CT with 5mm cuts in the treatment position, on a breast board, with both arms extended above their head. The organs at risk (heart, lungs) will be contoured on the CT scan.

The affected breast (with the index lesion) and associated lymphatic drainage will be treated according to the treating physician decision. The contralateral breast will be treated with 2 tangent fields, using 1.8-2 Gy/fx to a total dose of 50-50.4 Gy. The whole breast will be treated according to traditional guidelines and as described in the RTOG/NSABP B39 study. The heart should be completely blocked for left sided breasts, included lung tissue should be reduced to minimum. No overlapping field is allowed on the skin between the two breast fields in the midline. Maximal dose should not exceed 110%.

Follow up:

The treating physician will follow the patient every 2 weeks during the radiation treatment. Side effects will be scored and recorded in the patients chart according to the Common Terminology Criteria for Adverse Events v3.0.

Subsequent follow-up schedule according to the treating institution and ASCO guidelines. Patients will undergo annual mammogram and breasts US. Annual breasts MRI and bilateral salpingo-oophorectomy will be recommended.

Ipsilateral and contralateral breast cancer will be recorded and reported. Any subsequent malignancy other than breast cancer will be reported. Long-term radiation side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient diagnosed with stage I-III breast cancer (AJCC 6), undergoing breast irradiation as part of her adjuvant therapy.
2. The patient must be a carrier of a deleterious mutation in BRCA 1/2.
3. Age above 30 years.
4. The patient may receive any regimen of adjuvant chemotherapy, according to the treating physician. All cycles of chemotherapy must be completed at least 3 weeks prior to the start of radiation therapy.
5. The patient may be treated with hormonal therapy before, during or after study entry, according to the guidelines of her treating center.
6. The patient must have negative gadolinium based MRI of the contralateral breast, no more than 6 months prior to study entry.
7. The patient refused prophylactic contralateral mastectomy.
8. The patient is aware that subsequent breast cancer in the irradiated breast will probably mandate mastectomy.
9. The patient consent for contralateral prophylactic irradiation. -

Exclusion Criteria:

1. Metastatic breast cancer.
2. Previous irradiation of the breast or chest wall.
3. Pregnancy.
4. No concurrent chemotherapy is allowed
5. Patients with active connective tissue diseases are excluded due to the potential risk of significant radiotherapy toxicity.
6. Patients who are unable to lie on their back and raise their arms above their heads in the treatment planning position for radiotherapy are excluded -

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-03; Primary Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Rate of contralateral breast cancer in carrier patients that received prophylactic radiation to the contralateral breast compared with carrier patients that did not receive that treatment. | 15 years
  To compare the rate of contralateral breast cancer in carrier patients that received prophylactic radiation to the contralateral breast to the rate in carrier patients that did not receive that treatment

SECONDARY OUTCOMES:
Short and long term adverse effects of prophylactic contralateral breast irradiation. | 15 years
factors that influence patient's choice of treatment | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Ella Evron, MD, Study Director — Assaf-Harofeh Medical Center
Locations (1):
- Assaf-Harofeh Medical Center, Zerrifin, Israel

REFERENCES:
- [Background] Pierce LJ, Levin AM, Rebbeck TR, Ben-David MA, Friedman E, Solin LJ, Harris EE, Gaffney DK, Haffty BG, Dawson LA, Narod SA, Olivotto IA, Eisen A, Whelan TJ, Olopade OI, Isaacs C, Merajver SD, Wong JS, Garber JE, Weber BL. Ten-year multi-institutional results of breast-conserving surgery and radiotherapy in BRCA1/2-associated stage I/II breast cancer. J Clin Oncol. 2006 Jun 1;24(16):2437-43. doi: 10.1200/JCO.2005.02.7888. Epub 2006 Apr 24. PMID 16636335
- [Background] Metcalfe K, Lynch HT, Ghadirian P, Tung N, Olivotto I, Warner E, Olopade OI, Eisen A, Weber B, McLennan J, Sun P, Foulkes WD, Narod SA. Contralateral breast cancer in BRCA1 and BRCA2 mutation carriers. J Clin Oncol. 2004 Jun 15;22(12):2328-35. doi: 10.1200/JCO.2004.04.033. PMID 15197194
- [Derived] Evron E, Goldberg H, Ben-David MA, Corn BW. Participation in a Novel Trial Assessing Prophylactic Breast Irradiation: The Importance of Input From the Radiation Oncologist. Int J Radiat Oncol Biol Phys. 2019 Nov 15;105(4):792-794. doi: 10.1016/j.ijrobp.2019.08.004. Epub 2019 Aug 10. No abstract available. PMID 31408668
- [Derived] Evron E, Ben-David AM, Goldberg H, Fried G, Kaufman B, Catane R, Pfeffer MR, Geffen DB, Chernobelsky P, Karni T, Abdah-Bortnyak R, Rosengarten O, Matceyevsky D, Inbar M, Kuten A, Corn BW. Prophylactic irradiation to the contralateral breast for BRCA mutation carriers with early-stage breast cancer. Ann Oncol. 2019 Mar 1;30(3):412-417. doi: 10.1093/annonc/mdy515. PMID 30475942